CLINICAL TRIAL: NCT05392218
Title: Behavioral Intervention to Promote Healthy Lifestyle Behaviors: A Feasibility Randomized Controlled Trial
Brief Title: Behavioral Intervention to Promote Healthy Lifestyle Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Shaima Alothman, Associate Researcher, Clinical Assistant Professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-0142
Record Dates: First submitted 2022-05-09; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Health-Related Behavior
MeSH Terms: conditions — Health Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motivational interviewing (Experimental)
  Interventions: Behavioral: motivational interviewing
- attention group (Sham Comparator)
  Interventions: Behavioral: general health education

INTERVENTIONS:
Behavioral: motivational interviewing — consisted of six sessions (twice each week) up to 30 minutes of individual sessions. Each session contained a different component and topic that included substance abuse, physical activity, healthy sleep, stress management, nutrition and social support. The components in order were randomized for each participant.
  Arms: motivational interviewing
Behavioral: general health education — rceived the same amount of virtual session equivalent to MI form. However, the structure of the sessions consisted of brief advice to promote healthy lifestyle delivered by different therapists
  Arms: attention group

SUMMARY:
in this study to "the investigators aim to improve lifestyle behaviors through behavioral interventions. Participants will be assigned to one of two groups. both groups will be asked to complete online survey before and after a 6 virtual session (twice weekly)

DETAILED DESCRIPTION:
Participants were randomly assigned into two groups (motivational interviewing intervention or attention group), using a (1:1) computer-generated randomization program (www.graphpad.com).

motivational interviewing intervention: Each session contained a different component and topic that included substance abuse, physical activity, healthy sleep, stress management, nutrition and social support. The components in order were randomized for each participant. Interviews were conducted using a video meeting platform (Zoom Video Communications Inc., 2016); with both video and audio function enabled while, participants were giving the choice to refuse video calls should they desire. Alternative session delivery method, such as phone calls were used and documented based on participant request.

attention group: received the same amount of virtual session equivalent to MI form. However, the structure of the sessions consisted of brief advice to promote healthy lifestyle delivered by different therapists. The therapist firmly and clearly discussed general lifestyle health topics and provided educational materials during each session

ELIGIBILITY:
Inclusion Criteria:

* living in Saudi Arabia with stay home advisory
* speak Arabic

Exclusion Criteria:

* confirmed or suspected COVID-19 diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
recruitment rate - descriptive | immediately after the intervention
  reported as the number of participants' consented divide by the number of people that were invited to participate
retention rates - descriptive | immediately after the intervention
  reported as the number of participants completing all study sessions
session duration - descriptive | immediately after the intervention
  reported as the average session time for intervention group or attention group

SECONDARY OUTCOMES:
physical activity and sedentary behavior - questionnaire | outcome measure was assessed at baseline and within 7 days from the last study session
  measured via Global Physical Activity. physical activity level was calculated based on responses. sedentary behavior was reported as average sitting time per day.
psychosocial distress - questionnaire | outcome measure was assessed at baseline and within 7 days from the last study session
  via Kessler Psychological Distress Scale (K10). score range from 10 to 50 and higher scores reflecting higher psychological distress
sleep - questionnaire | outcome measure was assessed at baseline and within 7 days from the last study session
  via Pittsburgh Sleep Quality Index (PSQI). score ranges from 0 to 21. Poor sleepers have ≥ 5 scores as a cut-off global score
dietary habits - questionnaire | outcome measure was assessed at baseline and within 7 days from the last study session
  via food frequency questionnaire (FFQ). data reported as count
social support - questionnaire | outcome measure was assessed at baseline and within 7 days from the last study session
  via Medical Outcomes Study (MOS) Social Support Survey. This tool contains 19 questions, and higher score indicates more social support
fear of COVID-19 - questionnaire | outcome measure was assessed at baseline and within 7 days from the last study session
  via Fear of COVID-19 Scale (FCV-19S). score ranging from 7 to 35. The higher score indicates a higher fear of COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Alothman SA, Alshehri MM, Almasud AA, Aljubairi MS, Alrashed I, Abu Shaphe M, Alghannam AF. Virtual Behavioral Intervention to Promote Healthy Lifestyle Behaviors: A Feasibility RCT during COVID-19 Pandemic. Healthcare (Basel). 2022 Dec 28;11(1):91. doi: 10.3390/healthcare11010091. PMID 36611550